CLINICAL TRIAL: NCT00613951
Title: A 16 Week Randomised, Open Labelled, 3-armed, Parallel Group, Treat-to-target Trial Comparing Twice Daily (BID) Injections of SIAC 30 (B), SIAC 45 (B) and NovoMix®30, All in Combination With Metformin in Subjects With Type 2 Diabetes Failing on OAD Treatment
Brief Title: Comparison of Two NN5401 Formulations Versus Biphasic Insulin Aspart 30, All in Combination With Metformin in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-1792; 2007-002462-35 (EudraCT Number)
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Results first posted 2015-12-01 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination; insulin aspart, insulin aspart protamine drug combination 30:70; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SIAC 30 (B) (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart; Drug: metformin
- SIAC 45 (B) (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart; Drug: metformin
- BIAsp 30 (Active Comparator)
  Interventions: Drug: biphasic insulin aspart; Drug: metformin

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Formulation B: Treat-to-target dose titration scheme, injection s.c., twice daily
  Arms: SIAC 30 (B)
Drug: insulin degludec/insulin aspart — Formulation B: Treat-to-target dose titration scheme, injection s.c., twice daily
  Arms: SIAC 45 (B)
Drug: biphasic insulin aspart — Treat-to-target dose titration scheme, injection s.c., twice daily
  Arms: BIAsp 30
Drug: metformin — Tablets, 1500-2000 mg/daily

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare two NN5401 (Soluble Insulin Analogue Combination [SIAC], insulin degludec/insulin aspart) formulations with each other and with biphasic insulin aspart 30, all in combination with metformin in insulin naive subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject.)
* Insulin naïve type 2 diabetes subjects (as diagnosed clinically) for at least 3 months (no previous insulin treatment or previous short term insulin treatment maximum 14 days within the last 3 months)
* Treatment with one or two oral anti-diabetic drugs (OADs): metformin, sulfonylurea, other insulin secretagogue (e.g. repaglinide, nateglinide), alpha-glucosidase inhibitors for at least 2 months at a stable maximally tolerated dose or at least half maximally allowed dose according to locally approved summary of product characteristics (SPC)
* HbA1c, 7.0-11.0 % (both inclusive)
* Body Mass Index (BMI), 25.0-37.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Metformin contraindication according to local practice
* Thiazolidinedione (TZD) treatment within previous 3 months prior to Visit 1
* Any systemic treatment with products, which in the investigator's opinion could interfere with glucose or lipid metabolism (e.g. systemic corticosteroids) within 3 months prior to randomisation
* Subject has a clinically significant, active (during the past 12 months) disease of the gastrointestinal, pulmonary, neurological, genitourinary, or haematological system (except for conditions associated with type 2 diabetes) that, in the opinion of the investigator, may confound the results of the trial or pose additional risk in administering trial product

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (31):
- Finland (4):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Kuopio
  - Novo Nordisk Investigational Site, Lahti
  - Novo Nordisk Investigational Site, Pori
- France (7):
  - Novo Nordisk Investigational Site, Bar-le-Duc
  - Novo Nordisk Investigational Site, Grenoble
  - Novo Nordisk Investigational Site, Hayange
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Nanterre
  - Novo Nordisk Investigational Site, Nevers
  - Novo Nordisk Investigational Site, Pointe à Pitre
- Germany (7):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Pirna
  - Novo Nordisk Investigational Site, Riesa
  - Novo Nordisk Investigational Site, Saarbrücken
  - Novo Nordisk Investigational Site, Saint Ingbert
  - Novo Nordisk Investigational Site, Völklingen
  - Novo Nordisk Investigational Site, Wangen
- Poland (8):
  - Novo Nordisk Investigational Site, Bydgoszcz
  - Novo Nordisk Investigational Site, Gniewkowo
  - Novo Nordisk Investigational Site, Nysa
  - Novo Nordisk Investigational Site, Płock
  - Novo Nordisk Investigational Site, Szczecin
  - Novo Nordisk Investigational Site, Tychy
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw
- Spain (5):
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Granada
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, San Juan

REFERENCES:
- [Result] Niskanen L, Leiter LA, Franek E, Weng J, Damci T, Munoz-Torres M, Donnet JP, Endahl L, Skjoth TV, Vaag A. Comparison of a soluble co-formulation of insulin degludec/insulin aspart vs biphasic insulin aspart 30 in type 2 diabetes: a randomised trial. Eur J Endocrinol. 2012 Aug;167(2):287-94. doi: 10.1530/EJE-12-0293. Epub 2012 Jun 1. PMID 22660026
- [Result] Ma Z, Parkner T, Christiansen JS, Laursen T. IDegAsp: a novel soluble insulin analogs combination. Expert Opin Biol Ther. 2012 Nov;12(11):1533-40. doi: 10.1517/14712598.2012.722203. Epub 2012 Sep 4. PMID 22946603
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 27 sites in 5 countries: Finland (4), France (4), Germany (6), Poland (9) and Spain (4).
Pre-assignment Details: Subjects underwent a run-in period of up to 3 weeks (including 1-week maintenance period) where metformin was up-titrated to 1500 or 2000 mg/day. Subjects who tolerated metformin dose for a week and had fasting plasma glucose ≥ 7.5 mmol/L were randomised to SIAC 30 (B), SIAC 45 (B) or BIAsp 30 twice daily.
Groups:
- SIAC 30 (B): Soluble Insulin Analogue Combination 30 (SIAC 30, 70 volume percent insulin degludec, 600 nmol/ml and 30 volume percent insulin aspart, 600 nmol/ml [1 dosing unit = 6 nmol]); formulation B) was given subcutaneously twice daily before breakfast and dinner in combination with at least 1500 mg metformin (tablets) for 16 weeks. Insulin doses were individually adjusted.
- SIAC 45 (B): Soluble Insulin Analogue Combination 45 (SIAC 45, 55 volume percent insulin degludec, 600 nmol/ml and 45 volume percent insulin aspart, 600 nmol/ml [1 dosing unit = 6 nmol]); formulation B) was given subcutaneously twice daily before breakfast and dinner in combination with at least 1500 mg metformin (tablets) for 16 weeks. Insulin doses were individually adjusted.
- BIAsp 30: Biphasic insulin aspart 30 (BIAsp 30) was given subcutaneously twice daily before breakfast and dinner in combination with at least 1500 mg metformin (tablets) for 16 weeks. Insulin doses were individually adjusted.
Period: Overall Study
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | BIAsp 30
Started | 61 | 59 | 62
Exposed | 60 (One subject withdrew prior to exposure to trial drug) | 59 | 62
Completed | 54 | 54 | 57
Not Completed | 7 | 5 | 5
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Lack of Efficacy | 0 | 1 | 1
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Unclassified | 5 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | BIAsp 30 | Total
Number analyzed (Participants) | 61 | 59 | 62 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (8.5) | 60.5 (8.9) | 59.7 (8.0) | 59.6 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 30 | 23 | 85
  Male | 29 | 29 | 39 | 97
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.5 (1.2) | 8.5 (0.9) | 8.6 (1.0) | 8.5 (1.1)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 11.4 (2.7) | 11.8 (2.9) | 11.7 (3.1) | 11.6 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline in HbA1c after 16 weeks of treatment
Time Frame: Week 0, Week 16
Population: The full analysis set (FAS) included all randomised subjects and missing data was imputed using last observation carried forward (LOCF). HbA1c values were missing for 2 subjects, hence did not contribute to the analysis
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | BIAsp 30
Number analyzed (Participants) | 60 | 58 | 62
percentage of glycosylated haemoglobin | -1.79 (1.11) | -1.87 (0.91) | -1.84 (0.93)

2. Secondary Outcome: Mean of 9-point Self Measured Plasma Glucose Profile (SMPG)
Description: Estimate of the overall mean of SMPG after 16 weeks of treatment. Plasma glucose measured: before breakfast, 120 minutes after start of breakfast, before lunch, 120 minutes after start of lunch, before dinner, 120 minutes after start of dinner, before bedtime, at 4 am and before breakfast.
Time Frame: Week 16
Population: The full analysis set (FAS) included all randomised subjects and missing data was imputed using last observation carried forward (LOCF). For 2 subjects, mean SMPG values were missing.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | BIAsp 30
Number analyzed (Participants) | 60 | 58 | 62
mmol/L | 7.52 (0.27) | 7.44 (0.28) | 7.52 (0.27)

3. Secondary Outcome: Rate of Major and Minor Hypoglycaemic Episodes
Description: Observed rate of major and minor hypoglycaemic episodes per 100 patient years of exposure (PYE). Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: Week 0 to Week 16 + 5 days follow up
Population: The full analysis set (FAS) included all randomised subjects.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | BIAsp 30
Number analyzed (Participants) | 61 | 59 | 62
Episodes/100 years of patient exposure
  Major | 0 | 0 | 0
  Minor | 287 | 679 | 730

4. Secondary Outcome: Rate of Nocturnal Major and Minor Hypoglycaemic Episodes
Description: Rate of nocturnal major and minor hypoglycaemic episodes per 100 patient years of exposure (PYE). Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose below 3.1 mmol/L. Episodes were defined as nocturnal if the time of onset was between 23:00 (included) and 05:59 (included).
Time Frame: Week 0 to Week 16 + 5 days follow up
Population: The full analysis set (FAS) included all randomised subjects.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | BIAsp 30
Number analyzed (Participants) | 61 | 59 | 62
Episodes/100 years of patient exposure
  Major | 0 | 0 | 0
  Minor | 39 | 79 | 108

5. Secondary Outcome: Rate of Treatment Emergent Adverse Events (AEs)
Description: Corresponds to rate of AEs per 100 patient years of exposure. Severity assessed by investigator. Mild: no or transient symptoms, no interference with subject's daily activities. Moderate: marked symptoms, moderate interference with subject's daily activities. Severe: considerable interference with subject's daily activities, unacceptable. Serious AE: AE that at any dose results in any of the following: death, a life-threatening experience, in-subject hospitalization/prolongation of existing hospitalisation, persistent/significant disability/incapacity/congenital anomaly/birth defect.
Time Frame: Week 0 to Week 16 + 5 days follow up
Population: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Events/100 years of patient exposure
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | BIAsp 30
Number analyzed (Participants) | 60 | 59 | 62
Events/100 years of patient exposure
  Adverse events (AEs) | 298 | 545 | 379
  Serious AEs | 0 | 0 | 11
  Severe AEs | 0 | 0 | 5
  Moderate AEs | 56 | 67 | 38
  Mild AEs | 242 | 477 | 335
  Fatal AEs | 0 | 0 | 5

6. Secondary Outcome: Laboratory Safety Parameters (Biochemistry): Alanine Aminotransferase (ALAT)
Description: Laboratory values at screening (Week -4) and at Week 16
Time Frame: Week -4, Week 16
Population: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator. For 2 subjects the laboratory values were missing at week -4. From the SAS, 54 (SIAC 30), 57 (SIAC 45) and 53 (BIAsp 30) subjects contributed to the analysis at week 16.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | BIAsp 30
Number analyzed (Participants) | 60 | 59 | 62
IU/L
  Week -4, N=60, 57, 62 | 33.0 (16.6) | 31.4 (16.0) | 36.9 (23.4)
  Week 16, N=54, 57, 53 | 22.9 (9.2) | 22.5 (11.1) | 23.6 (11.3)

7. Secondary Outcome: Laboratory Safety Parameters (Biochemistry): Aspartate Aminotransferase (ASAT)
Description: Laboratory values at screening (Week -4) and at Week 16
Time Frame: Week -4, Week 16
Population: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator. For 3 subjects the laboratory values were missing at week -4. From the SAS, 54 (SIAC 30), 57 (SIAC 45) and 53 (BIAsp 30) subjects contributed to the analysis at week 16.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | BIAsp 30
Number analyzed (Participants) | 60 | 59 | 62
IU/L
  Week -4, N=60, 56, 62 | 23.6 (11.2) | 25.2 (12.0) | 26.4 (16.1)
  Week 16, N=54, 57, 53 | 22.6 (8.7) | 22.9 (11.4) | 23.1 (11.2)

8. Secondary Outcome: Laboratory Safety Parameters (Biochemistry): Serum Creatinine
Description: Laboratory values at screening (Week -4) and at Week 16
Time Frame: Week -4, Week 16
Population: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator. For 2 subjects the laboratory values were missing at week -4. From the SAS, 56 (SIAC 30), 57 (SIAC 45) and 56 (BIAsp 30) subjects contributed to the analysis at week 16.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | BIAsp 30
Number analyzed (Participants) | 60 | 59 | 62
umol/L
  Week -4, N=60, 57, 62 | 72.7 (14.0) | 75.8 (14.8) | 74.8 (14.1)
  Week 16, N=56, 57, 56 | 73.6 (13.2) | 76.3 (16.1) | 78.1 (15.5)

9. Secondary Outcome: Vital Signs: Diastolic Blood Pressure (BP)
Description: Values at baseline (Week 0) and at Week 16
Time Frame: Week 0, Week 16
Population: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator. From the SAS, 58 (SIAC 30), 56 (SIAC 45) and 58 (BIAsp 30) subjects contributed to the analysis at week 16.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | BIAsp 30
Number analyzed (Participants) | 60 | 59 | 62
mmHg
  Week 0 (Baseline), N=60, 59, 62 | 80 (9) | 81 (10) | 81 (11)
  Week 16, N=58, 56, 58 | 78 (9) | 79 (10) | 76 (9)

10. Secondary Outcome: Vital Signs: Systolic Blood Pressure (BP)
Description: Values at baseline (Week 0) and at Week 16
Time Frame: Week 0, Week 16
Population: The safety analysis set includes all subjects who received at least one dose of the investigational product or its comparator. From the SAS, 58 (SIAC 30), 56 (SIAC 45) and 58 (BIAsp 30) subjects contributed to the analysis at week 16.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | BIAsp 30
Number analyzed (Participants) | 60 | 59 | 62
mmHg
  Week 0 (Baseline), N=60, 59, 62 | 134 (15) | 138 (18) | 137 (18)
  Week 16, N=58, 56, 58 | 128 (13) | 135 (17) | 133 (15)

11. Secondary Outcome: Vital Signs: Pulse
Description: Values at baseline (Week 0) and at Week 16
Time Frame: Week 0, Week 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | BIAsp 30
Number analyzed (Participants) | 60 | 59 | 62
beats/minute
  Week 0 (Baseline), N=60, 59, 62 | 74 (10) | 76 (8) | 75 (8)
  Week 16, N=58, 56, 58 | 73 (10) | 73 (8) | 77 (9)

12. Secondary Outcome: Physical Examination
Description: Physical examination was performed at screening (week -4), and after 8 and 16 weeks of treatment. If any new findings or deterioration in previous findings were observed during the trial, these were recorded as AEs and are therefore not presented separately as no analysis was performed.
Time Frame: Week -4, Week 8, Week 16
Arm/Group | BIAsp 30 | SIAC 30 (B) | SIAC 45 (B)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 16 weeks + 5 days follow up
Description: The safety analysis set included all subjects with exposure information of at least one dose of randomised trial medication.
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | BIAsp 30
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/59 | 2/62
Other Adverse Events (participants affected / at risk) | 14/60 | 13/59 | 13/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SIAC 30 (B) (N=60) | SIAC 45 (B) (N=59) | BIAsp 30 (N=62)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SIAC 30 (B) (N=60) | SIAC 45 (B) (N=59) | BIAsp 30 (N=62)
Oedema peripheral (General disorders) | 0 (0) | 4 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 8 (9) | 4 (4) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (7) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (4) | 4 (7)
Headache (Nervous system disorders) | 6 (10) | 5 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.